CLINICAL TRIAL: NCT05826340
Title: A 3-arm Randomised Parallel Group Superiority Trial to Investigate the Efficacy of Graded Loading and Return to Sport or Pain Guided Activity, Versus Rest or on Symptom and Disease Severity in Patients With Osgood Schlatter
Brief Title: Getting Kids With Osgood Schlatter Back to Performing Without Pain
Acronym: QUICKRETURNOSD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aalborg University (Other)
Responsible Party: Principal Investigator, Sinead Holden, Investigator, Aalborg University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Quick Return OSD 001; N-20210052 (Other: VEK RN)
Record Dates: First submitted 2023-01-26; First posted 2023-04-24 (Actual); Last update posted 2023-04-24 (Actual); Status verified 2023-04

CONDITIONS: Osgood-Schlatter Disease
Keywords: Growth; Adolescent; Musculoskeletal; Pain; Osteochondrosis
MeSH Terms: conditions — Osteochondrosis; Pain

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Tailored loading (Experimental): Participants will be provided with a 5-stage return to sport tool, which gradually increases sports intensity and knee loading. In addition, they are to perform a progressive exercise program at home to increase lower extremity strength and prepare them for the demands of sport. Participants will begin at a starting point in the five stages based on their current symptoms and self reported sports related disability, and given guidance on how to progress / regress their loading within the five stage framework
  Interventions: Behavioral: Tailored progressive loading and return to sport
- Pain within acitvity limits (Experimental): Participants will be advised to participate in sport/exercise to the extent that pain allows. They will not be restriced full from sport but will be instructed how to use a pain moritoring tool to help monitor pain and balance the amount of activities in which they can participate.
  Interventions: Behavioral: Pain guided activity
- Rest until pain subsides (No Intervention): Participants will be provided advice on rest for a minimum of four weeks or until pain subsides

INTERVENTIONS:
Behavioral: Tailored progressive loading and return to sport — Participants will undergo a 5-stage progressive return to sport tool.
  Other Names: Progressive return to sport
  Arms: Tailored loading
Behavioral: Pain guided activity — Participants will be provided on information on how to guide activity based on pain response.
  Arms: Pain within acitvity limits

SUMMARY:
The goal of this trial is to compare graded return to sport, or pain guided activity to rest in youth with Osgood Schlatter. The main objectives are:

- to assess the graded return to sport, or pain guided activity on symptoms (pain and function) at six months compared to rest

The secondary objectives are to assess the impact of progressive return to sport or pain guided activity on:

* Muscle strength and performance
* Anterior knee pain provocation
* Sports participation
* Physical activity

The exploratory objectives are to assess the impact of progressive return to sport on ultrasound imaging characteristics of OSD.

DETAILED DESCRIPTION:
Osgood Schlatter disease (OSD) affects 10% of adolescents aged 9-15. This makes it the most common knee pain condition in this age group. OSD is considered an overuse injury, common in highly sports active adolescents. It is considered an apophyseal injury of the tibial tuberosity, the site of attachment of the patellar tendon onto the tibia. Repetitive forces exerted on tissues without allowing for recovery can cause pain and/or tissue damage at the site of attachment onto the weak developing apophyseal cartilage which is thought to be a susceptible injury before the apophysis is fully matured. Characteristics such as cartilage swelling, and associated tendon changes (including thickening of the patellar tendon and increased doppler activity) have been documented.

Despite narrative reviews recommending conservative management, there is a complete lack of clinical research evaluating the different recommendations, which range from passive interventions, such as rest/activity limitation, to more active approaches including strength exercises for the lower extremity. We have developed a new progressive return to sport intervention approach which has been piloted in adolescents with OSD. The targeted intervention aims to balance recovery, and graded loading in a guided return to sport paradigm The goal is to help support adolescents manage pain, and guide return to sport & function.

There is a need to test other potential conservative interventions which have yet to be examined in a randomised manner. Multi-arm trials allow more treatments to be assessed than a standard two arm trial. This makes this design simpler, quicker and cheaper than running multiple two arm trials, which will produce contemporaneous results for all treatments. This is relevant in the context of OSD, where none of the conservative recommendations have been evaluated. Despite rest being advocated, it may be possible to allow adolescents to participants to participate in sports to the extent that pain allows (pain guided activity). This may be beneficial, given the social and health consequences of complete withdrawal from sport. We therefore aim to evaluate both the progressive return to sport paradigm and pain guided activity in a 3-armed randomised trial, compared to advice to rest and withdrawal from sports.

ELIGIBILITY:
Inclusion Criteria:

- Children/adolescents (male and female) aged 8-16 years

* Diagnosis of OSD based on clinical examination including localised pain at the tibial tuberosity (the insertion of the patellar tendon onto the shin) that increases by palpation, and pain during resisted isometric knee extension.
* Ability to understand and the willingness to provide consent

Exclusion Criteria:

* Any other diagnosable knee pathology, patellar instability, and patellofemoral instability.
* Previous knee surgery
* Habitual patella subluxation
* Clinical suspicion of meniscal lesion
* Previous neurologic, musculoskeletal or mental illnesses
* Other chronic conditions that may affect the involved musculoloskeletal/connective tissues and treatment (autoimmune, metabolic disorders, diabetes, etc.)
* Lack of ability to cooperate

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 144 (Estimated)
Dates: Start 2023-01-26 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | 6 months
  Pain intensity will be captured using a visual analogue scale (VAS) ranging from 0cm (no pain) to 10cm (worst pain imaginable) where participants are asked to rate their worth pain in the previous week.
Sports related function | 6 months
  The patient reported questionnaire Knee Injury and Osteoarthritis Outcome Score (KOOS) contains five separate subscales. We will use the KOOS-Child Sport/Rec subscale to assess sports related function.The scale ranges from 0-100, with higher scores indicating better outcomes

SECONDARY OUTCOMES:
Health related quality of life | 3 months, 6 months, 12 months
  Health related quality of life will be measured by the youth version of the European Quality of Life 5 Dimensions (EQ-5D-Y) at baseline, 3months, 6 months and 12months. The index score ranges from 0-1, with 1 indicating full health.
Muscle strength and performance | 6 months
  Isometric knee extension torque, hip abduction, and hip extension torque will be measured using a handheld dynamometer. Participants will perform three maximal effort contractions. Results will be averaged and normalised to body weight and lever length.
  Lower limb power will be conducted by asking the participants to perform single leg vertical and horizontal jumps.
Sports participation | 3months, 6months, 12 months
  Adolescents will report their weekly sports volume (expressed in hours per week).
Return to sport | 3months, 6months, 12 months
  In case of any absence from sport, the time to return to sport (i.e. duration of absence) will be documented.
Objective physical activity | 6 months
  Participants will be provided with an Actigraph monitor for two weeks to objectively measure physical activity (time spent in moderate to vigorous physical activity and sedentary time at 6 months follow-up. The specific model used will be the wGT3X- BT actigraphy device (ActiGraphCorp, Pensacola, FL), which is a compact, wrist- worn, battery-powered, CE marked device that captures and records continuous, high resolution physical activity and sleep/wake information.
Pain severity during palpation | 6 months
  Numeric rating scale ranging from 0, no pain to 10 worst imaginable pain) in response to palpation of the tibial tuberosity.
Pain severity during knee loading | 6 months
  Numeric rating scale ranging from 0, no pain to 10 worst imaginable pain) in response to the anterior knee pain provocation (AKPP). Participants will be asked to complete a single leg squat to about 60 degrees of knee flexion and hold the position for 30 seconds. Pain will be recorded at the end of 30 seconds.
Global rating of change | 3 months, 6 months, 12 months
  Self-reported recovery on a 7-point Likert scale, ranging from much better, to much worse.
Pain intensity | 3 months, 12 months
  Pain intensity will be captured using a visual analogue scale (VAS) ranging from 0cm (no pain) to 10cm (worst pain imaginable) where participants are asked to rate their worth pain in the previous week.
Sports related function | 3 months, 12 months
  The patient reported questionnaire Knee Injury and Osteoarthritis Outcome Score (KOOS)[22] contains five separate subscales. We will use the KOOS-Child Sport/Rec subscale to assess sports related function. This scale ranges from 0-100 with higher scores reflecting better outcomes

OTHER OUTCOMES:
OSD ultrasound staging according to DeFlaviis | 6 months
  Ultrasound scans of the knee will be used at baseline and six months to evaluate OSD ultrasound classification according to DeFlaviis (no changes, cartilage swelling, cartilage swelling plus bony changes, associated bursitis, associated tendonopathy).
Ulstrasound characteristics: neovascularisation | 6 months
  Ultrasound scans of the knee will be used at baseline and six months to evaluate neovascularisation in the tendon and apophysis. This will be done by evaluating the presence of positive Doppler signal.
Ulstrasound characteristics: tendon thickness | 6 months
  Ultrasound scans of the knee will be used at baseline and six months to evaluate tendon thickness at the distal patellar tendon. To determine distal thickness, a transversal scan taken 1cm from TT attachment will be used.
Patient satisfaction | 3months ,6 months, 12 months
  Patient satisfaction with the results of the treatment will be asked on a 5-point Likert scale ranging from very satisfied to very unsatisfied.

CONTACTS AND LOCATIONS:
Overall Officials: Sinead Holden, PhD, Principal Investigator — Aalborg University; Michael S Rathleff, Dr. Med, Principal Investigator — Aalborg University; Jens Olesen, Principal Investigator — Centre for Almen Medicin ved Aalborg Universitet
Locations (1):
- Research Unit for General Practice in Aalborg, Aalborg, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Data will be managed according to the FAIR principles (findable, accessible, inter-operable and reproducible). Meta-data will be uploaded to Open Science framework with restrictions and terms for accessing the anonymised data according for research purposes, where appropriate.
Supporting Information: Study Protocol
Time Frame: Anticipated after study completion and publication